CLINICAL TRIAL: NCT02935530
Title: Effectiveness and Safety of Thromboprophylaxis After Surgery for Gynecologic Malignancy in China
Brief Title: Thromboprophylaxis After Surgery for Gynecologic Malignancy in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ding Ma, Director of the department of Obstetrics and Gynecology, Tongji Hospital, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VTE-01
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Gynecologic Neoplasms; Venous Thromboembolism; Low Molecular Weight Heparin; Argatroban
MeSH Terms: conditions — Genital Neoplasms, Female; Venous Thromboembolism | interventions — Heparin, Low-Molecular-Weight; argatroban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- s-LMWH (Experimental): 2125 I.U. subcutaneous injection for 5-10 days
  Interventions: Drug: s-LMWH
- LMWH (Active Comparator): 4250 I.U. subcutaneous injection for 5-10 days
  Interventions: Drug: LMWH
- Argatroban (Experimental): 20mg, injection for 5-10 days
  Interventions: Drug: Argatroban

INTERVENTIONS:
Drug: s-LMWH — 2125KU, subcutaneous injection of 5-10 days
  Arms: s-LMWH
Drug: LMWH — 4250KU, subcutaneous injection of 5-10 days
  Arms: LMWH
Drug: Argatroban — 20mg, injection for 5-10 days
  Arms: Argatroban

SUMMARY:
Venous thromboembolism (VTE) is an important cause of post-operative morbidity and mortality in women undergoing surgery for gynecologic malignancies. Although the benefit of thromboprophylaxis in reduction of post-operative VTE events after surgery for gynecologic cancers has been well documented around the world, the evidence for Chinese women is rare. The investigators designed this prospective and randomized study to assess the benefit of pharmacologic prophylaxis for patients received surgical treatment for gynecologic malignancies in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients of ovarian cancer, cervix cancer or endometrial cancer;
* Age ≤ 70 years; female, Chinese women;
* Initial treatment is surgery;
* Laboratory tests: WBC ≥ 4×10(9)/L, NEU ≥ 2×10(9)/L, PLT ≥ 100×10(9)/L, serum bilirubin ≤ 1.5 times the upper limit of normal, transaminase ≤ 1.5 times the upper limit of normal, BUN, Cr ≤ normal
* No prior pharmacologic prophylaxis;
* Provide written informed consent.

Exclusion Criteria:

* PLT ≤ 75×10(9)/L
* Vascular injury
* History of thrombosis
* Liver and kidney dysfunction
* Concurrently participating in other clinical trials
* Unable or unwilling to sign informed consents;
* Unable or unwilling to abide by protocol.

Ages: 16 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
VTE rate | 30-days from the date of operation

SECONDARY OUTCOMES:
Bleeding rate | 30-days from the date of operation
Infection rate | 30-days from the date of operation

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, M.D., Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No